CLINICAL TRIAL: NCT00107003
Title: A Biomarker and Phase II Study of GW572016 in Recurrent Malignant Glioma
Brief Title: GW572016 to Treat Recurrent Malignant Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 050134; 05-C-0134; NCT00103129 (obsolete NCT alias)
Record Dates: First submitted 2005-04-02; First posted 2005-04-04 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2012-11-30

CONDITIONS: Glioma; Brain Tumor; Glioblastoma Multiforme; GBM; Gliosarcoma; GS
Keywords: Brain; Tumor; Surgery; Therapy; Trial; Brain Tumor; Glioblastoma Multiforme; GBM; Gliosarcoma; GS
MeSH Terms: conditions — Glioma; Brain Neoplasms; Glioblastoma; Gliosarcoma; Neoplasms | interventions — Lapatinib; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: lapatinib ditosylate
Procedure: Adjuvant therapy
Procedure: Conventional surgery
Procedure: Neoadjuvant therapy

SUMMARY:
This study will examine whether an experimental drug called GW572016 can delay tumor growth in patients with glioblastoma multiforme (GMB, a malignant brain tumor). GW572016 is believed to affect cancer cell function by interfering with the internal signaling needed for the cancer to grow. The study will also determine whether the presence of specific proteins in the tumor can predict what effects GW572016 will have on the tumor.

Patients 18 years of age and older with GMB whose brain tumor does not respond to standard medical treatment and who can undergo surgery for their tumor may be eligible for this study. Candidates are screened with a physical examination and neurocognitive examination, blood tests, electrocardiogram (EKG), echocardiogram (ultrasound test of heart function) or MUGA scan (nuclear medicine test of heart function), magnetic resonance imaging (MRI) of the head, and computed tomography (CT) of the head. CT uses x-rays and MRI uses a magnetic field and radio waves to show brain structure.

Participants undergo the following tests and procedures:

* MRI and blood tests before surgery.
* Surgery to remove the brain tumor.
* Follow-up MRIs every 8 weeks after surgery.
* Follow-up echocardiograms or MUGA scans every 8 weeks after surgery.
* GW572016 treatment starting 7-10 days before surgery and continuing until the patient or doctor decides it is in the patient's best interest to stop it or until the tumor worsens. (The drug is stopped temporarily for surgery and a healing period after surgery.)
* Blood tests every 2 weeks to evaluate the effects of GW572016 on the body.
* Blood test before the first GW572016 treatment and at the time of surgery to assess the effect of the drug on the cells and to determine how much drug is present in the blood at the time of surgery.

Participants are followed in clinic at least monthly while taking GW572016. While on treatment they keep a diary documenting their daily treatments. The diary is collected at the monthly follow-up exams. After the treatment ends, patients are contacted periodically by the research staff for the rest of their lives to follow the long-term effects of the study.

DETAILED DESCRIPTION:
Background:

- One of the most critical challenges facing glioblastoma translational research is developing ways to predict, based on a patient's biopsy, which targeted inhibitor is most likely to provide benefit. The studies outlined in this proposal are designed to determine which glioblastoma patients are most likely to benefit from GW572106, and may provide a blueprint for analyzing promising new pathway inhibitors in the future. We anticipate that these studies will serve as the basis for biological endpoint based trials in the future. Thus, the overall goal is to evaluate the efficacy of GW572016 in the treatment of recurrent malignant gliomas in patients who are candidates for re-resection.

Objective:

* Determine the 6-month progression-free survival rate for patients with recurrent or progressive glioblastoma treated with GW572016.
* Determine whether GW572016 inhibits the phosphorylation of its cellular targets EGFR and HER2, and the downstream PI3K-AKT and RAS-ERK signaling pathways in glioblastoma patients in vivo.
* Determine tumor concentrations of GW572016.
* Assess overall progression free survival and safety.

Eligibility:

* Patients with histologically proven intracranial tumors to include only glioblastoma multiforme (GBM) and Gliosarcoma (GS). Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a GBM is made.
* Patients must be candidates for surgical re-resection (total, or sub-total) in order to be eligible for this study. Following surgery, a scan should be done no later than 96 hours
* Patients may be on a non-enzyme-inducing anti-epileptic drugs (Non-EIAED's). They may not be on EIAED's. If previously on an EIAED, patient must be off of it for two weeks prior to initiation of pre-operative drug.

Design:

* A Pre-Treatment blood sample (10ml) will be obtained in all patients for genotyping
* Pre- Operative: GW572016 will be administered at a starting dose of 750 mg orally BID daily on an outpatient basis for 7-10 days. (This range is to allow flexibility for planning surgery). GW572016 will be continued up to and including the evening before surgery.
* At the time of surgery 10ml of blood will be collected in EDTA containing tubes for pharmacodynamic analysis
* Treatment may be instituted postoperatively as soon as patients have recovered from effects of surgery and demonstrated wound healing. Treatment with GW572016 post-operatively should start no later than 28 days after surgery. GW572016 will be administered at a starting dose of 750 mg orally BID daily on an outpatient basis. GW572016 will be administered continuously; however, for the purposes of protocol evaluations, a cycle will be defined as 28 days.

ELIGIBILITY:
* INCLUSION CRITERIA (General):

Patients with histologically proven intracranial tumors to include only glioblastoma multiforme (GBM) and Gliosarcoma (GS). Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a GBM is made.

Unstained slides (at least 5, but prefer 10) or 1 tissue block must be available from at least one prior surgery. If available, frozen tissue is also requested from earlier surgeries.

Patients must be candidates for surgical re-resection (total, or sub-total) in order to be eligible for this study. Following surgery, a scan should be done no later than 96 hours.

Patients may be on a non-enzyme-inducing anti-epileptic drugs (Non-EIAED's). They may not be on EIAED's. If previously on an EIAED, patient must be off of it for two weeks prior to initiation of pre-operative drug.

Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan (within 42 days of registration).

All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information. Patients must be registered in the NABTC database prior to treatment with study drug.

Patients must be greater than or equal to 18 years old, and with a life expectancy greater than 8 weeks.

Patients must have a Karnofsky performance status of greater than or equal to 60.

Patients must have recovered from the toxic effects of prior therapy and at least 28 days from any investigational agent, 28 days from prior cytotoxic therapy, 28 days from radiation, 14 days from vincristine, 42 days from nitrosoureas, 21 days from procarbazine administration, and 7 days from non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.

Patients must have adequate bone marrow function (WBC greater than or equal to 3,000/microl, ANC greater than or equal to 1,500/mm(3), platelet count of greater than or equal to 100,000/mm(3), and hemoglobin greater than or equal to 10 gm/dl), adequate liver function (SGOT and bilirubin less than 2.5 times ULN), and adequate renal function (creatinine less than 1.5 mg/dL before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.

Patients must have shown unequivocal evidence for tumor progression by MRI or CT scan. Stable dose of steroids is not mandated for this study. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.

Patients must have failed prior radiation therapy.

Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or Thallium scanning, MR spectroscopy or surgical documentation of disease.

Patients may have had treatment for no more than 2 prior relapses. Relapse is defined as progression following initial therapy (i.e. radiation+/- chemo [which includes gliadel wafers] if that was used as initial therapy). The intent therefore is that patients had no more than 3 prior therapies (initial and treatment for 2 relapses). If the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered as 1 relapse. For patients who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse.

Eligibility to restart drug post-op.

Patients must agree to practice adequate contraception. Women of childbearing potential must have a negative B-HCG pregnancy test documented within 7 days prior to registration.

EXCLUSION CRITERIA (General):

Patients may not be on any medications listed in section 3.2.1

Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.

Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years are ineligible.

Patients must not have active infection or serious intercurrent medical illness.

Women of childbearing potential must not be pregnant/breast feeding. Patients must not be pregnant because no studies with this drug have been performed to evaluate safety.

HIV-Positive patients receiving combination anti-retroviral therapy are excluded from the study due to possible retro-viral drug interactions.

Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.

Patients must not have received prior therapy with Signal transduction inhibitors (e.g. ZD1839, OSI-774, R115777)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-03-30; Primary Completion 2007-12-05 (Actual); Study Completion 2012-11-30 (Actual)

PRIMARY OUTCOMES:
Determine 6-month progression-free survival of patients undergoing surgery for recurrent progressive glioblastoma multiforme or gliosarcoma treated with lapatinib.

CONTACTS AND LOCATIONS:
Overall Officials: Teri N Kreisl, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Burgess AW, Cho HS, Eigenbrot C, Ferguson KM, Garrett TP, Leahy DJ, Lemmon MA, Sliwkowski MX, Ward CW, Yokoyama S. An open-and-shut case? Recent insights into the activation of EGF/ErbB receptors. Mol Cell. 2003 Sep;12(3):541-52. doi: 10.1016/s1097-2765(03)00350-2. PMID 14527402
- [Background] Choe G, Park JK, Jouben-Steele L, Kremen TJ, Liau LM, Vinters HV, Cloughesy TF, Mischel PS. Active matrix metalloproteinase 9 expression is associated with primary glioblastoma subtype. Clin Cancer Res. 2002 Sep;8(9):2894-901. PMID 12231534
- [Background] Hendriks BS, Opresko LK, Wiley HS, Lauffenburger D. Quantitative analysis of HER2-mediated effects on HER2 and epidermal growth factor receptor endocytosis: distribution of homo- and heterodimers depends on relative HER2 levels. J Biol Chem. 2003 Jun 27;278(26):23343-51. doi: 10.1074/jbc.M300477200. Epub 2003 Apr 9. PMID 12686539